CLINICAL TRIAL: NCT00000693
Title: Suppression of Cytomegalovirus Retinitis Utilizing High Dose Intravenous Acyclovir and Oral Zidovudine in Patients With AIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 070; 11044 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Cytomegalovirus Retinitis; HIV Infections
Keywords: Retinitis; Drug Evaluation; Drug Therapy, Combination; Cytomegalovirus Infections; Acyclovir; Acquired Immunodeficiency Syndrome; Zidovudine
MeSH Terms: conditions — Cytomegalovirus Retinitis; HIV Infections; Retinitis; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome | interventions — Zidovudine; Acyclovir

INTERVENTIONS:
Drug: Zidovudine
Drug: Acyclovir

SUMMARY:
To study the use of acyclovir (ACV) and zidovudine (AZT) in the treatment of cytomegalovirus (CMV) retinitis in patients with AIDS who would otherwise be treated with ganciclovir (DHPG) alone.

CMV retinitis is one of the most common opportunistic infections in patients with AIDS. DHPG is at present the only drug available for widespread compassionate use in the United States. Although most patients respond to treatment with DHPG, the medication does not cure the infection. Most patients will have a relapse and will require retreatment with DHPG. Because of the large relapse rate, most people treated for CMV retinitis are placed on continuous treatment with DHPG. There are two major problems associated with ongoing use of DHPG: 1) The development of a low white blood cell (WBC) count (leukopenia) which is a known side effect of the drug; and 2) the increased risk for leukopenia when DHPG is given together with AZT, the only antiviral drug currently available for the treatment of HIV infection. Therefore, patients cannot take both AZT and DHPG at the same time because the bone marrow toxicity is made much more severe when the drugs are given together. This has resulted in the difficult decision as to whether to forgo potential life-extending therapy with AZT in order to preserve sight. An effective treatment for CMV retinitis is needed that will allow the patient to also take AZT. ACV is presently the drug of choice for severe herpes virus infections. It has been shown to be effective in suppressing severe CMV disease in patients who have received bone marrow transplants.

DETAILED DESCRIPTION:
CMV retinitis is one of the most common opportunistic infections in patients with AIDS. DHPG is at present the only drug available for widespread compassionate use in the United States. Although most patients respond to treatment with DHPG, the medication does not cure the infection. Most patients will have a relapse and will require retreatment with DHPG. Because of the large relapse rate, most people treated for CMV retinitis are placed on continuous treatment with DHPG. There are two major problems associated with ongoing use of DHPG: 1) The development of a low white blood cell (WBC) count (leukopenia) which is a known side effect of the drug; and 2) the increased risk for leukopenia when DHPG is given together with AZT, the only antiviral drug currently available for the treatment of HIV infection. Therefore, patients cannot take both AZT and DHPG at the same time because the bone marrow toxicity is made much more severe when the drugs are given together. This has resulted in the difficult decision as to whether to forgo potential life-extending therapy with AZT in order to preserve sight. An effective treatment for CMV retinitis is needed that will allow the patient to also take AZT. ACV is presently the drug of choice for severe herpes virus infections. It has been shown to be effective in suppressing severe CMV disease in patients who have received bone marrow transplants.

Patients receive ACV intravenously and AZT orally for 12 weeks. Tolerance of the combined administration of ACV and AZT is monitored. AMENDED: AZT dose lowered and inclusion of concurrent medication expanded.

ELIGIBILITY:
Inclusion Criteria

Prior Medication:

Required:

* Patients must have successfully completed remission induction therapy with ganciclovir (minimum of 14 days of therapy) for acute cytomegalovirus (CMV) retinitis within the preceding 48 hours. Patients who show no evidence of progressive disease are considered to have met criteria for successful induction.

Amended to allow:

* Investigational triazoles.
* Human recombinant erythropoietin (Eprex).
* Other investigational non-antiviral therapies offered through treatment IND.

Patients must:

* Have HIV infection as determined by a commercially licensed ELISA test confirmed by a licensed Western blot
* Have salvageable vision (corrected acuity of 20/100 or better) in at least one eye.
* Be capable of signing an informed consent.

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Known or suspected allergy to one of the study medications.
* Inability to maintain adequate hydration status.

Concurrent Medication:

Excluded:

* Concurrent therapy with nephrotoxic agents.
* Systemic therapy for another opportunistic infection.
* Systemic prophylaxis for Pneumocystis carinii pneumonia (PCP).
* Probenecid.
* Patients are advised that validity of this trial may be jeopardized by use of other potentially antiviral or immunomodulating treatments.

Patients with the following are excluded:

* Known or suspected allergy to one of the study medications.
* Inability to maintain adequate hydration status.

Prior Medication:

Excluded within 2 weeks of study entry:

* Steroids.
* Cytotoxic or immunosuppressive drugs.
* Investigational agents. (Amended to now allow these.) Immunomodulatory drugs (except ganciclovir).

Prior Treatment:

Excluded within 2 weeks of study entry:

* Radiotherapy.

Risk Behavior:

Excluded:

* History of unreliable drug intake and inability to cooperate in the testing procedures. Unwilling or unable to give informed consent or unwilling to sign approved consent form.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25
Dates: Study Completion 1992-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: HA Kessler, Study Chair; CA Benson, Study Chair
Locations (2):
- United States (2):
  - Northwestern Univ Med School, Chicago, Illinois
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois

REFERENCES:
- [Background] Sha BE, Benson CA, Deutsch TA, Urbanski PA, Phair JP, Kessler HA. Suppression of cytomegalovirus retinitis in persons with AIDS with high-dose intravenous acyclovir. J Infect Dis. 1991 Oct;164(4):777-80. doi: 10.1093/infdis/164.4.777. PMID 1654361